CLINICAL TRIAL: NCT01280955
Title: A Phase I/II Study: Enhancing Donor Hematopoietic Cell Engraftment With Plerixafor in Myeloablative Allogeneic Hematopoietic Cell Transplantation
Brief Title: Donor Enhancement With Plerixafor Post Myeloablative Allogeneic Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mitchell Horwitz, MD (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Mitchell Horwitz, MD, Assoc Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00024433
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Failure of Bone Marrow Graft
Keywords: Plerixafor and Allogeneic Myeloablative Stem Cell Transplant
MeSH Terms: interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant Recipients (Experimental): Transplant recipients from matched sibling donors and dual cord donors. Subjects will receive plerixafor at 240 ug/kg subcutaneously every other day beginning at day +2 after transplant until day +21 or engraftment occurs.
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Matched sibling or Dual Cord donor subjects will receive plerixafor at 240 ug/kg subcutaneously every other day beginning at day +2 after transplant until day +21 or engraftment occurs.
  Other Names: AMD3100; Mozobil

SUMMARY:
This phase I/II clinical trial will test the safety and the efficacy of post transplant administration of plerixafor in enhancing hematological recovery in humans. Patients who are appropriate candidates for myeloablative allogeneic stem cell transplantation from an HLA-matched sibling, matched unrelated donor or umbilical cord blood are eligible for enrollment. The investigators plan to enroll a total of 50 patients for this study (30 patients with HLA-matched sibling or matched unrelated donor transplant, and 20 patients with umbilical cord blood transplant). During phase I study, a small number of patients (3-6 patients from each group) will be enrolled to determine the safety of post transplant administration of plerixafor. Patients will receive plerixafor given at 240 µg/kg subcutaneously every other day beginning at day +2 after transplant until day +21 or engraftment. Limiting toxicities are defined as primary or secondary graft failure, plerixafor-related severe premature ventricular arrhythmia or death. If safety criteria are met from the investigators phase I study, the investigators will proceed with phase II study to determine the efficacy of post transplant administration of plerixafor in enhancing haematological recovery. The experimental aspect of this study is the use of plerixafor and all other aspects of care will be in line with the standard of care. Both Phase I and Phase II patients will be combined for efficacy analysis, and data collected from this study will be compared with the investigators historical control. The results from this study will set the stage and provide the justification for a larger phase 3 trial.

DETAILED DESCRIPTION:
Recruitment to this trial will be stratified by donor type as HLA (human leukocyte antigen) matched sibling, matched unrelated donor or umbilical cord blood. Patients will be conditioned with a myeloablative regimen such as, but not limited to, total body irradiation and cyclophosphamide. The donor stem cell grafts will come from mobilized peripheral blood of 8/8 or 7/8 HLA-identical family members, 8/8 (HLA A, B, C, DRBeta1) allele-level matched unrelated donors, or dual umbilical cord blood grafts with at least 4 of 6 HLA matching at HLA A and B (low resolution) and DRBeta1 (at high resolution). The target CD34+ cell dose will be 5 X 10(6)/kg recipient ideal body weight. For HLA matched sibling or matched unrelated donor (MUD) transplants, all patients will receive a minimum of 2 X 10(6) CD 24+ cells/kg. For cord blood transplants, each unit will contain a minimum total nucleated cell count of of 1.5 X 10(7)/kg. Post-transplant GVHD (graft versus host disease) prophylaxis will be given per institutional standard.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years.
* 8/8 or 7/8 HLA-identical matched sibling OR Allele level 8/8 (HLA-A, B, C, DR Beta1)matched unrelated donor or 4/6 or better HLA matched cord blood.
* Patients with high risk hematologic malignancies who are appropriate candidates for a myeloablative allogeneic stem cell transplantation.
* Patients with a history of CNS disease must have been treated and have no active CNS disease at the time of protocol treatment.
* ECOG performance status < or equal to 2
* Patients must have adequate function of other organ systems as measured by:
* Creatinine clearance (by Cockcroft Gault equation) > or equal to 30ml/min. Hepatic transaminases (ALT/AST) < or equal to 4 x normal, bilirubin < or equal to 2.0 mg/dl.
* Pulmonary function tests demonstrating FVC and FEV1 of > or equal to 50% of predicted for age and DLCO > or equal to 50% of predicted.
* Ejection fraction of > or equal to 45% by echocardiogram, radionuclide scan or cardiac MRI.
* Patients must be HIV negative.
* Patients must not be pregnant.

Exclusion Criteria:

* Patients with > 5% blasts in bone marrow or peripheral circulation.
* Uncontrolled infection.
* Class III or IV angina as per NYHA criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Principal Investigator — Duke University; Saurabh Chhabra, MD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Green MM, Chao N, Chhabra S, Corbet K, Gasparetto C, Horwitz A, Li Z, Venkata JK, Long G, Mims A, Rizzieri D, Sarantopoulos S, Stuart R, Sung AD, Sullivan KM, Costa L, Horwitz M, Kang Y. Plerixafor (a CXCR4 antagonist) following myeloablative allogeneic hematopoietic stem cell transplantation enhances hematopoietic recovery. J Hematol Oncol. 2016 Aug 17;9(1):71. doi: 10.1186/s13045-016-0301-2. PMID 27535663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who are appropriate candidates for myeloablative allogeneic stem cell transplantation from an HLA-matched sibling, matched unrelated donor or umbilical cord blood are eligible for enrollment. The first subject was consented on 9/28/2011. The study closed to accrual on 5/27/2014.
Pre-assignment Details: 41 participants signed consent and 30 received transplant. 11 patients who signed consent were screen failures. Reasons patients did not receive transplant included lack of donor, insurance denial, too much disease, uncontrolled infection, class III or IV angina. 29 participants were used in results analysis because one participant withdrew.
Groups:
- Transplant Recipients: This arm includes transplant recipients from matched sibling donors and dual cord donors. Subjects will receive plerixafor at 240 ug/kg subcutaneously every other day beginning at day +2 after transplant until day +21 or engraftment occurs.
Period: Overall Study
Arm/Group | Transplant Recipients
Started | 30
Completed | 27
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline includes transplant recipients only and excludes 1 patient who withdrew from the study.
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Time to Neutrophil Recovery
Description: leukocytes > 500/ul on 2 consecutive days
Time Frame: 100 Days post Transplant
Population: Out of the 30 transplant recipients, one participant withdrew and was therefore not analyzed
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Transplant Recipients: This arm includes transplant recipients from matched sibling donors and dual cord blood donors. Subjects will receive plerixafor at 240 ug/kg subcutaneously every other day beginning at day +2 after transplant until day +21 or engraftment occurs.
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 29
days | 17 [16 to 18]

2. Primary Outcome: Time to Platelet Recovery
Description: platelet > 20,000/ul on 2 consecutive days
Time Frame: 100 Days Post Transplant
Population: Out of the 30 transplant recipients, one participant withdrew and was therefore not analyzed
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 29
days | 18 [15 to 22]

3. Primary Outcome: Plerixafor-associated Adverse Events
Time Frame: 100 Days Post Transplant
Population: Out of the 30 transplant recipients, one participant withdrew and was therefore not analyzed
Measure: Number; unit: number of adverse events
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 29
number of adverse events
  GI upset | 1
  nausea | 1
  diarrhea | 2
  fatigue | 1
  rash | 1
  pneumonia | 3
  bruising | 1

4. Secondary Outcome: Transplant-related Mortality
Time Frame: 100 Days Post Transplant
Population: Out of the 30 transplant recipients, one participant withdrew and was therefore not analyzed
Measure: Number; unit: participants
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 29
participants | 11

5. Secondary Outcome: Absolute Lymphocyte Count at Day 90
Description: Cell reconstitution - absolute lymphocyte count at day 90 post transplant.
Time Frame: 90 days
Population: the population includes all participants for which we have data at day 90
Measure: Median (Full Range); unit: number of lymphocytes
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 11
number of lymphocytes | 549 [209 to 2219]

6. Secondary Outcome: IL-12 at Day 30
Description: IL-12 at day 30; Interleukin 12 (IL-12) is an interleukin that is naturally produced by dendritic cells, macrophages, neutrophils, and human B-lymphoblastoid cells (NC-37) in response to antigenic stimulation.
Time Frame: 30 days
Population: the population includes all participants for which we have data at day 30
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 26
pg/mL | 40.7 [3.9 to 211.6]

7. Secondary Outcome: Participants Experiencing Grade II-IV Acute Graft Versus Host Disease
Description: We are reporting on the number of participants experiencing a grade II-IV acute graft versus host disease will be assessed weekly through Day 100 post transplant. Staging and grading of Acute GvHD is graded by pattern of organ involvement and clinical performance status using the Grading Index of Acute GvHD (Gluckman) and the Grading Index of Acute GVHD by the CIBMTR (Centers for International Blood and Marrow Transplant Research)
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 29
participants
  Grade 2 | 5
  Grade 3 | 5

8. Secondary Outcome: CD3+ Cell Count at Day 90
Description: Cell reconstitution - CD3+ cell count at day 90 post transplant. This is a marker for the function of your immune system.
Time Frame: 90 Days
Population: the population includes all participants for which we have data at day 90
Measure: Median (Full Range); unit: number of CD3+ cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 11
number of CD3+ cells | 655 [128 to 1656]

9. Secondary Outcome: CD4 Cell Count at Day 90
Description: CD4 cell count at Day 90; CD4+ T helper cells are white blood cells that are an essential part of the human immune system. They are often referred to as CD4 cells, T-helper cells or T4 cells.
Time Frame: 90 days
Population: The population includes subjects for which we have data at day 90.
Measure: Median (Full Range); unit: number of CD4 cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 11
number of CD4 cells | 180 [59 to 596]

10. Secondary Outcome: CD8 Cell Count at Day 90
Description: CD8 cell count at Day 90; CD8 (cluster of differentiation 8) is a transmembrane glycoprotein that serves as a co-receptor for the T cell receptor (TCR).
Time Frame: 90 days
Population: the population includes subjects for which we have data at day 90
Measure: Median (Full Range); unit: number of CD8 cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 11
number of CD8 cells | 172 [31 to 1209]

11. Secondary Outcome: NK Cell Count at Day 90
Description: NK cell count at Day 90;Natural killer cells or NK cells are a type of cytotoxic lymphocyte critical to the immune system.
Time Frame: 90 days
Population: the population includes subjects for which we have data at Day 90.
Measure: Median (Full Range); unit: number of NK cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 11
number of NK cells | 137 [42 to 495]

12. Secondary Outcome: B Cell Count at Day 90
Description: B cell count at Day 90; B cells, also known as B lymphocytes, are a type of white blood cell of the lymphocyte subtype and they function as part of the immune system.
Time Frame: 90 days
Population: the population includes subjects for which we have data at Day 90.
Measure: Median (Full Range); unit: number of B cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 11
number of B cells | 7 [0 to 128]

13. Secondary Outcome: IFN Gamma at Day 30
Description: IFN gamma at day 30; Interferon gamma (IFNγ) is a dimerized soluble cytokine that is the only member of the type II class of interferons which are important for immunity against infection.
Time Frame: 30 days
Population: the population includes subject for which we have data at Day 30.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 26
pg/mL | 8.6 [0 to 80.7]

14. Secondary Outcome: TNF-alpha at Day 30
Description: TNF-alpha at day 30; Tumor necrosis factor is a cell signaling protein (cytokine) involved in systemic inflammation and is one of the cytokines that make up the acute phase reaction. The primary role of TNF is in the regulation of immune cells.
Time Frame: 30 days
Population: the population includes subject for which we have data at Day 30.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 26
pg/mL | 146.5 [0 to 551.6]

15. Secondary Outcome: CD4 Cell Count at Day 30
Description: CD4 cell count at Day 30; CD4+ T helper cells are white blood cells that are an essential part of the human immune system. They are often referred to as CD4 cells, T-helper cells or T4 cells.
Time Frame: 30 days
Population: The population includes subjects for which we have data at day 30.
Measure: Median (Full Range); unit: number of CD4 cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 13
number of CD4 cells | 252 [75 to 552]

16. Secondary Outcome: CD4 Cell Count at Day 60
Description: CD4 cell count at Day 60; CD4+ T helper cells are white blood cells that are an essential part of the human immune system. They are often referred to as CD4 cells, T-helper cells or T4 cells.
Time Frame: 60 days
Population: The population includes subjects for which we have data at day 30.
Measure: Median (Full Range); unit: number of CD4 cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 6
number of CD4 cells | 220 [67 to 317]

17. Secondary Outcome: CD8 Cell Count at Day 30
Description: CD8 cell count at Day 30; CD8 (cluster of differentiation 8) is a transmembrane glycoprotein that serves as a co-receptor for the T cell receptor (TCR).
Time Frame: 30 days
Population: the population includes subjects for which we have data at day 30
Measure: Median (Full Range); unit: number of CD8 cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 13
number of CD8 cells | 255 [15 to 1766]

18. Secondary Outcome: CD8 Cell Count at Day 60
Description: CD8 cell count at Day 60; CD8 (cluster of differentiation 8) is a transmembrane glycoprotein that serves as a co-receptor for the T cell receptor (TCR).
Time Frame: 60 days
Population: the population includes subjects for which we have data at day 60
Measure: Median (Full Range); unit: number of CD8 cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 6
number of CD8 cells | 199 [92 to 609]

19. Secondary Outcome: NK Cell Count at Day 30
Description: NK cell count at Day 30;Natural killer cells or NK cells are a type of cytotoxic lymphocyte critical to the immune system.
Time Frame: 30 days
Population: the population includes subjects for which we have data at Day 30.
Measure: Median (Full Range); unit: number of NK cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 13
number of NK cells | 226 [22 to 376]

20. Secondary Outcome: NK Cell Count at Day 60
Description: NK cell count at Day 60;Natural killer cells or NK cells are a type of cytotoxic lymphocyte critical to the immune system.
Time Frame: 60 days
Population: the population includes subjects for which we have data at Day 60.
Measure: Median (Full Range); unit: number of NK cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 6
number of NK cells | 221 [33 to 315]

21. Secondary Outcome: B Cell Count at Day 30
Description: B cell count at Day 30; B cells, also known as B lymphocytes, are a type of white blood cell of the lymphocyte subtype and they function as part of the immune system.
Time Frame: 30 days
Population: the population includes subjects for which we have data at Day 30.
Measure: Median (Full Range); unit: number of B cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 13
number of B cells | 6 [1 to 42]

22. Secondary Outcome: B Cell Count at Day 60
Description: B cell count at Day 60; B cells, also known as B lymphocytes, are a type of white blood cell of the lymphocyte subtype and they function as part of the immune system.
Time Frame: 60 days
Population: the population includes subjects for which we have data at Day 60.
Measure: Median (Full Range); unit: number of B cells
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 6
number of B cells | 18 [0 to 158]

23. Secondary Outcome: IL-12 at Day 7
Description: IL-12 at day 7; Interleukin 12 (IL-12) is an interleukin that is naturally produced by dendritic cells, macrophages, neutrophils, and human B-lymphoblastoid cells (NC-37) in response to antigenic stimulation.
Time Frame: 7 days
Population: the population includes all participants for which we have data at day 7
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 28
pg/mL | 8.4 [2.4 to 90]

24. Secondary Outcome: IL-12 at Day 14
Description: IL-12 at day 14; Interleukin 12 (IL-12) is an interleukin that is naturally produced by dendritic cells, macrophages, neutrophils, and human B-lymphoblastoid cells (NC-37) in response to antigenic stimulation.
Time Frame: 14 days
Population: the population includes all participants for which we have data at day 14
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 27
pg/mL | 13.3 [0.9 to 222.1]

25. Secondary Outcome: IFN Gamma at Day 7
Description: IFN gamma at day 7; Interferon gamma (IFNγ) is a dimerized soluble cytokine that is the only member of the type II class of interferons which are important for immunity against infection.
Time Frame: 7 days
Population: the population includes subject for which we have data at Day 7.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 28
pg/mL | 3.9 [0 to 116.3]

26. Secondary Outcome: IFN Gamma at Day 14
Description: IFN gamma at day 14; Interferon gamma (IFNγ) is a dimerized soluble cytokine that is the only member of the type II class of interferons which are important for immunity against infection.
Time Frame: 14 days
Population: the population includes subject for which we have data at Day 14.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 27
pg/mL | 20.0 [0 to 243.5]

27. Secondary Outcome: TNF-alpha at Day 7
Description: TNF-alpha at day 7; Tumor necrosis factor is a cell signaling protein (cytokine) involved in systemic inflammation and is one of the cytokines that make up the acute phase reaction. The primary role of TNF is in the regulation of immune cells.
Time Frame: 7 days
Population: the population includes subject for which we have data at Day 7.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 28
pg/mL | 15.9 [0 to 162.6]

28. Secondary Outcome: TNF-alpha at Day 14
Description: TNF-alpha at day 14; Tumor necrosis factor is a cell signaling protein (cytokine) involved in systemic inflammation and is one of the cytokines that make up the acute phase reaction. The primary role of TNF is in the regulation of immune cells.
Time Frame: 14 days
Population: the population includes subject for which we have data at Day 14.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 27
pg/mL | 43.8 [0.9 to 190.6]

ADVERSE EVENTS:
Time Frame: adverse events are collected for 1 year post transplant
Description: Adverse Events were monitored for 29 transplant recipients
Groups:
- Transplant Recipients: This arm includes transplant recipients from matched sibling donors and dual cord blood donors. Subjects will receive plerixafor at 240 ug/kg subcutaneously every other day beginning at day +2 after transplant until day +21 or engraftment occurs.
  Adverse Events were monitored for 29 transplant recipients
Arm/Group | Transplant Recipients
Serious Adverse Events (participants affected / at risk) | 12/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant Recipients (N=29)
encephalitis (Infections and infestations) | 1 (1) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Brain (encephalitis, infectious)
death (General disorders) | 4 (4) — Death Not Associated with CTCAE term - Death NOS
pneumonia (Infections and infestations) | 1 (1) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Lung (pneumonia)
small bowel (NOS) (Infections and infestations) | 1 (1) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Small bowel NOS
death (General disorders) | 3 (3) — Death Not Associated with CTCAE term - Disease Progression NOS
death (General disorders) | 2 (2) — Death Not Associated with CTCAE term - Multi-Organ Failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant Recipients (N=29)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3 (4)
hypogammagloulinemia (Immune system disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 5 (7)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 2 (2)
presbyacusis (Hearing loss) (Nervous system disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (2)
Bladder spasms (Renal and urinary disorders) | 1 (1)
engraftment syndrome (Blood and lymphatic system disorders) | 2 (2)
anemia (Blood and lymphatic system disorders) | 1 (1)
pancytopenia (Blood and lymphatic system disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 1 (1)
relapsed disease (Blood and lymphatic system disorders) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 4 (4)
tacycardia (Cardiac disorders) | 7 (9)
Confusion (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
pyrexia (fever) (General disorders) | 6 (6)
fatigue (General disorders) | 1 (1)
frail appearance (General disorders) | 1 (2)
hyperthermia (overheating) (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 3 (3)
Dental: caries (General disorders) | 1 (1)
contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
groin irratation (Skin and subcutaneous tissue disorders) | 1 (1)
pallor (Skin and subcutaneous tissue disorders) | 1 (2)
erythema (Skin and subcutaneous tissue disorders) | 1 (2)
scratch marks (Skin and subcutaneous tissue disorders) | 1 (2)
purpuric lesion (Skin and subcutaneous tissue disorders) | 1 (1)
perianal lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 16 (24)
Dizziness (Nervous system disorders) | 3 (3)
keratoconjunctivitis (Dry Eye Syndrome) (Eye disorders) | 2 (2)
Dry mouth / salivary gland (xerostomia) (General disorders) | 1 (1)
xeroderma (Dry Skin) (Skin and subcutaneous tissue disorders) | 4 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Edema (Blood and lymphatic system disorders) | 13 (18)
Extremity-lower (gait / walking) (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 (11)
Febrile neutropenia (Infections and infestations) | 17 (19)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 5 (7)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
odynophagia (Gastrointestinal disorders) | 1 (1)
oropharyngeal erythema (Gastrointestinal disorders) | 7 (13)
pain - general body ache (General disorders) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hair Loss / Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 (4)
Hearing Loss (Ear and labyrinth disorders) | 1 (1)
Heartburn / dyspepsia (Gastrointestinal disorders) | 3 (4)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, pulmonary / upper respiratory (Blood and lymphatic system disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (5)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Febrile neutropenia (Infections and infestations) | 6 (8)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 9 (10)
viremia (Infections and infestations) | 10 (13)
rsv pneumonia (Infections and infestations) | 4 (4)
Infection with unknown ANC - Blood (Infections and infestations) | 2 (2)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with unknown ANC - Sinus (Infections and infestations) | 2 (3)
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 2 (3)
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1 (1)
Infection without febrile neutropenia (Infections and infestations) | 1 (3)
Insomnia (General disorders) | 5 (5)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 6 (6)
Mental status decrease (Nervous system disorders) | 3 (3)
Mood Alteration - Anxiety (Nervous system disorders) | 4 (4)
pain - headache (Nervous system disorders) | 3 (3)
Mucositis / Stomatitis (clinical exam) (Gastrointestinal disorders) | 28 (34)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 4 (5)
asthenia (Musculoskeletal and connective tissue disorders) | 6 (10)
Musculoskeletal / Soft Tissue injury (Musculoskeletal and connective tissue disorders) | 4 (6)
Nasal cavity / paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Respiratory, thoracic and mediastinal disorders) | 15 (25)
Neurology (Nervous system disorders) | 1 (3)
fall (Nervous system disorders) | 1 (1)
lethargy (Nervous system disorders) | 1 (1)
peripheral neuropathy (Nervous system disorders) | 2 (2)
Neutrophils / granulocytes (ANC / AGC) (Blood and lymphatic system disorders) | 1 (1)
subconjunctivial hemorrhage (Eye disorders) | 1 (2)
rheum (crusty eye) (Eye disorders) | 2 (4)
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 8 (10)
Pain - Back (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Chest / thorax NOS (Cardiac disorders) | 1 (1)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain - Head / headache (Nervous system disorders) | 6 (9)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain- groin (Musculoskeletal and connective tissue disorders) | 5 (8)
Pain - Ovulatory (Reproductive system and breast disorders) | 1 (1)
Pain - Throat / pharynx / larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
platelets (Blood and lymphatic system disorders) | 3 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis / pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Potassium, serum-low (hypokalemia) (Musculoskeletal and connective tissue disorders) | 3 (6)
Pruritus / itching (Skin and subcutaneous tissue disorders) | 2 (4)
Pulmonary / Upper Respiratory infiltrates (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Rash / desquamation (Skin and subcutaneous tissue disorders) | 13 (19)
Rash: acne / acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
hematuria (Renal and urinary disorders) | 8 (14)
Rigors / chills (General disorders) | 2 (3)
Sinus Tachycardia (Cardiac disorders) | 8 (10)
Taste Alteration (dysgeusia) (Metabolism and nutrition disorders) | 3 (3)
Thrombosis / embolism (vascular access-related) (Vascular disorders) | 3 (3)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (3)
polyuria (Urinary frequency / urgency) (Renal and urinary disorders) | 2 (2)
Vision - blurred vision (Eye disorders) | 1 (1)
photophobia (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (26)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (1)
Weight gain (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was limited to recipients of matched adult donor grafts

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No